CLINICAL TRIAL: NCT00815581
Title: Comparison of Photorefraction With Cycloautorefraction and Cycloretinoscopy at Emam Hosein Medical Centre in 2008-2009
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 8728
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2008-12

CONDITIONS: Amblyopia
Keywords: children between 1 to 10 years old; amblyopy
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- photorefraction (Other)
  Interventions: Device: photorefraction,cycloautorefraction,cycloretinoscopy

INTERVENTIONS:
Device: photorefraction,cycloautorefraction,cycloretinoscopy

SUMMARY:
Screening of refractory defect is one of major reason for amblyopy. Photorefraction is a new method with some advantages in treatment of this problem. In this study the investigators are going to compare the results of this surgery in children between 1 to 10 years old with cycloautorefraction in children above 3 years old.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopy
* Children between 1 to 10 years old

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Locations (1):
- Ophtalmic Research Centre, Tehran, Tehran Province, Iran